CLINICAL TRIAL: NCT01195636
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, and Systemic Exposure of Topical XPF-002 in Subjects With Postherpetic Neuralgia
Brief Title: A Crossover Study to Evaluate the Safety, Tolerability and Efficacy of XPF-002 in Subjects With Postherpetic Neuralgia (PHN)
Acronym: XEN402
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-002-201
Record Dates: First submitted 2010-08-31; First posted 2010-09-06 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Postherpetic Neuralgia
Keywords: Pain from Shingles, PHN, Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XPF-002 (Experimental)
  Interventions: Drug: XPF-002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XPF-002 — Twice daily application of XPF-002 ointment which contains 8% of the XPF-002 active ingredient
  Arms: XPF-002
Drug: Placebo — Twice daily application of Placebo ointment
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine if XPF-002 is safe and effective for the treatment of pain in subjects with Postherpetic Neuralgia

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years (inclusive);
* Males or females of non-childbearing potential (ie, 12 months or more of spontaneous amenorrhea, bilateral oophorectomy at least 6 months prior to randomization, hysterectomy with bilateral oophorectomy at least 6 months prior to randomization, or for females over 50 years of age, hysterectomy without bilateral oophorectomy at least 6 months prior to randomization);
* Male subjects with sexual partners of childbearing potential must agree to use contraception (abstinence, birth control pills, rings or patches, diaphragm and spermicide, intrauterine device, condom and vaginal spermicide, surgical sterilization, vasectomy, progestin implant or injection);
* Persistent pain for more than 6 months from the appearance of herpes zoster rash that is not located on the face, above the scalp hairline, or in proximity to mucous membranes;
* Diagnosis of PHN;
* Persistent neuropathic pain that involves at least 1 dermatome and covering no more than 400 cm2;
* Mean daily pain intensity score in the target area of greater than or equal to 4 on an 11-point Likert NRS for a minimum of 4 days during the single-blind, placebo run-in period;
* Subject agrees to take only the protocol-defined rescue medication as prescribed;
* Intact skin over the painful area to be treated; and
* Able and willing to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Subject with systemic disease that would put him/her at an additional risk or limit his/her ability to participate in the study in the opinion of the investigator;
* Creatinine clearance less than 30 mL/min;
* Subject with known history of human immunodeficiency virus, hepatitis C, or hepatitis B;
* Malignancy other than basal cell carcinoma and carcinoma in situ within the past 2 years;
* Subject with history of serious mental illness or psychiatric illness such as dementia, depression, or schizophrenia, that will limit his/her ability to comply with study procedures;
* Subject who is unable to apply, or have a care giver apply, study ointment to the area of most painful skin segments, BID, once within 2 hours of waking and once in the evening after dinner;
* Subject with known sensitivity to topical products;
* Subject with active herpes zoster lesions or dermatitis;
* Other severe or chronic pain that may impair the self-assessment of the pain due to PHN;
* Treatment with local anesthetic in the last 2 weeks or nerve blocks within the last 30 days;
* Subject who is taking any opioid medications to treat his/her PHN pain and is unable to washout of these medications for the duration of the study;
* Subject who is taking any prohibited medication and is unable to washout of these treatments for the duration of the study;
* Subject who is taking more than 2 permitted concomitant medications for the treatment of PHN and is unable to washout of all but 2 of these treatments for the duration of the study;
* Subject who is taking any local prescription or non-prescription therapy (lidocaine patch, transcutaneous electrical nerve stimulation, etc.) and is unable to washout of these treatments for the duration of the study;
* Subject who has used Qutenza® patches in the 90 days prior to screening or has used other capsaicin preparations on a daily basis in the 90 days prior to screening;
* Subject who has participated in more than 1 other topical study for pain and more than 3 other PHN clinical studies;
* Pregnant or lactating females;
* Subject who has an active history of alcohol or drug abuse;
* Subject who has participated in any other investigational study within 60 days prior to screening;
* Subject who is employed by the Sponsor, study staff, and their families; or
* Subject who has any condition that would make him/her, in the opinion of the investigator or Sponsor, unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Jonesboro, Arkansas
  - Lomita, California
  - Westlake Village, California
  - Bradenton, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Lexington, Kentucky
  - Bay City, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Hartsdale, New York
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Austin, Texas
  - Houston, Texas
  - Sugar Land, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- XPF-002 First, Then Placebo: In the first intervention period XPF-002 ointment (8% strength) was applied twice daily for 3 weeks. After a washout period, Placebo ointment was applied twice daily for 3 weeks in the second intervention period.
- Placebo First, Then XPF-002: In the first intervention period Placebo ointment was applied twice daily for 3 weeks. After a washout period, XPF-002 ointment (8% strength) was applied twice daily for 3 weeks in the second intervention period.
Period: First Intervention (3 Weeks)
Arm/Group | XPF-002 First, Then Placebo | Placebo First, Then XPF-002
Started | 35 | 35
Received at Least 1 Dose of Drug | 33 | 35
Completed | 30 | 32
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout Period (2 Weeks)
Arm/Group | XPF-002 First, Then Placebo | Placebo First, Then XPF-002
Started | 30 | 32
Completed | 28 | 29
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Period: Second Intervention (3 Weeks)
Arm/Group | XPF-002 First, Then Placebo | Placebo First, Then XPF-002
Started | 28 | 29
Completed | 27 | 27
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- XPF-002 First, Then Placebo: XPF-002 ointment applied twice daily for 3 weeks followed by Placebo ointment applied twice daily for 3 weeks (after a washout period)
- Placebo First, Then XPF-002: Placebo ointment applied twice daily for 3 weeks followed by XPF-002 ointment applied twice daily for 3 weeks (after a washout period)
- Total: Total of all reporting groups
Arm/Group | XPF-002 First, Then Placebo | Placebo First, Then XPF-002 | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 23 | 18 | 41
  >=65 years | 11 | 17 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.58) | 63.1 (9.73) | 60.7 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Pain Score From Baseline to Week 3 (With LOCF)
Description: Subjects recorded their pain scores 4 times each day (using an 11-point Likert numerical rating scale (NRS); 0-10, where 0 = no pain and 10 = worst pain imaginable). An average (mean) daily pain score was calculated.
  This measurement is the 'Change in mean daily pain score from baseline between the 3rd week of XPF-002 treatment and the 3rd week of placebo treatment for each subject'. Any missing mean daily pain scores were imputed using last observation carried forward (LOCF).
  The reduction in pain on each treatment compared to baseline is reported as a negative number. A larger negative number, indicates a greater reduction in pain. (A positive number would indicate pain was increased compared to baseline.)
Time Frame: 3 weeks
Population: The Efficacy Evaluable Population was used for this analysis. This population includes randomised subjects who recorded both baseline and post-baseline data in both treatment periods. The maximum number of subjects who could contribute to this population is 57.
  Last Observation Carried Forward (LOCF) was used to impute any missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- XPF-002: XPF-002: 8% strength ointment, applied twice daily for 3 weeks in either the first intervention period or second intervention period.
- Placebo: Placebo: Vehicle only ointment, applied twice daily for 3 weeks in either first intervention period or second intervention period.
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 56 | 56
units on a scale | -0.94 [-1.30 to -0.58] | -0.97 [-1.33 to -0.61]

2. Secondary Outcome: Change in Mean Daily Pain Score From Baseline to Week 1
Description: Subjects recorded their pain scores 4 times each day (using an 11-point Likert numerical rating scale (NRS); 0-10, where 0 = no pain and 10 = worst pain imaginable). An average (mean) daily pain score was calculated.
  This measurement is the 'Change in mean daily pain score from baseline between the 1st week of XPF-002 treatment and the 1st week of placebo treatment for each subject'. Missing data were not imputed.
  The reduction in pain on each treatment compared to baseline is reported as a negative number. A larger negative number, indicates a greater reduction in pain. (A positive number would indicate pain was increased compared to baseline.)
Time Frame: 1 week
Population: The Efficacy Evaluable Population was used for this analysis. This population includes randomised subjects who recorded both baseline and post-baseline data in both treatment periods.
  Missing data were not imputed. Only subjects who recorded sufficient pain scores in each treatment period were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 54 | 54
units on a scale | -0.42 [-0.73 to -0.11] | -0.55 [-0.86 to -0.24]

3. Secondary Outcome: Change in Mean Daily Pain Score From Baseline to Week 2
Description: Subjects recorded their pain scores 4 times each day (using an 11-point Likert numerical rating scale (NRS); 0-10, where 0 = no pain and 10 = worst pain imaginable). An average (mean) daily pain score was calculated.
  This measurement is the 'Change in mean daily pain score from baseline between the 2nd week of XPF-002 treatment and the 2nd week of placebo treatment for each subject'. Missing data were not imputed.
  The reduction in pain on each treatment compared to baseline is reported as a negative number. A larger negative number, indicates a greater reduction in pain. (A positive number would indicate pain was increased compared to baseline.)
Time Frame: 2 week
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 55 | 55
units on a scale | -0.74 [-1.07 to -0.41] | -0.70 [-1.03 to -0.37]

4. Secondary Outcome: Change in Mean Daily Pain Score From Baseline to Week 3
Description: Subjects recorded their pain scores 4 times each day (using an 11-point Likert numerical rating scale (NRS); 0-10, where 0 = no pain and 10 = worst pain imaginable). An average (mean) daily pain score was calculated.
  This measurement is the 'Change in mean daily pain score from baseline between the 3rd week of XPF-002 treatment and the 3rd week of placebo treatment for each subject'. Missing data were not imputed.
  The reduction in pain on each treatment compared to baseline is reported as a negative number. A larger negative number, indicates a greater reduction in pain. (A positive number would indicate pain was increased compared to baseline.)
Time Frame: 3 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 52 | 52
units on a scale | -0.96 [-1.33 to -0.58] | -0.96 [-1.34 to -0.59]

5. Secondary Outcome: Proportion of Subjects Achieving at Least a 1 Point Improvement in Mean Daily Pain Score (Measured Using the 11-point Likert NRS) From Baseline to Week 3 on XPF-002 Compared to Placebo
Description: Subjects recorded their pain scores 4 times each day (using an 11-point Likert numerical rating scale (NRS); 0-10, where 0 = no pain and 10 = worst pain imaginable). An average (mean) daily pain score was calculated.
Time Frame: 3 Weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 52 | 52
participants | 22 | 19

6. Secondary Outcome: Proportion of Subjects Achieving 50% Improvement in Mean Daily Pain Score From Baseline to Week 3 on XPF-002 Treatment Compared to Placebo Treatment
Time Frame: 3 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 52 | 52
participants | 15 | 6

7. Secondary Outcome: Proportion of Subjects Achieving 30% Improvement in Mean Daily Pain Score From Baseline to Week 3 on XPF-002 Treatment Compared to Placebo Treatment
Time Frame: 3 Weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 52 | 52
participants | 21 | 12

8. Secondary Outcome: Proportion of Subjects Using Rescue Analgesic Medications During XPF-002 Treatment Compared to Placebo Treatment
Time Frame: 3 Weeks
Measure: Number; unit: participants
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 57 | 57
participants | 38 | 40

9. Secondary Outcome: Change in Overall Neuropathic Pain Symptom Inventory (NPSI) From Baseline to Week 3 (With LOCF)
Description: Subjects completed the NPSI questionaire at various timepoints during the study. An overall NPSI score (the sum of 10 quantitative responses, each scored 0-10, max score = 100) was calculated each time the NPSI questionaire was completed.
  This measurement is the 'Change in Neuropathic Pain Symptom Inventory (NPSI) score from baseline between the 3rd week of XPF-002 treatment and the 3rd week of placebo treatment for each subject. If the NPSI score for Week 3 was missing, the last value from within the same treatment period was used (ie last observation carried forward (LOCF)).
  The reduction in NPSI on each treatment compared to baseline is reported as a negative number. A larger negative number, indicates a greater reduction in neuropathic pain symptoms. (A positive number would indicate neuropathic pain symptoms were increased compared to baseline.)
Time Frame: 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 53 | 53
units on a scale | -6.7 (16.28) | -6.1 (13.51)

10. Secondary Outcome: Change in Daily Sleep Interference Scale (DSIS) From Baseline to Week 3 of XPF-002 Treatment Compared to Week 3 of Placebo Treatment (With LOCF)
Description: Subjects recorded their sleep interference scores each morning for the previous night's sleep (using an 11-point Likert numerical rating scale (NRS); 0-10, where 0 = no interference with sleep and 10 = pain completely interfered with sleep). A daily sleep interference score was calculated.
  This measurement is the 'Change in DSIS score from baseline between the 3rd week of XPF-002 treatment and the 3rd week of placebo treatment for each subject'. Any missing scores were imputed using last observation carried forward (LOCF).
  The reduction in DSIS on each treatment compared to baseline is reported as a negative number. A larger negative number, indicates a greater reduction in sleep interference due to pain. (A positive number would indicate sleep interference due to pain was increased compared to baseline.)
Time Frame: 3 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | XPF-002 | Placebo
Number analyzed (Participants) | 53 | 53
units on a scale | -0.81 [-1.21 to -0.41] | -0.84 [-1.24 to -0.43]

ADVERSE EVENTS:
Arm/Group | XPF-002 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/62 | 1/63
Other Adverse Events (participants affected / at risk) | 12/62 | 17/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XPF-002 (N=62) | Placebo (N=63)
Tooth abcess (Infections and infestations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XPF-002 (N=62) | Placebo (N=63)
Application site pain (General disorders) | 2 | 10
Application site pruritus (General disorders) | 2 | 8
Application site exfoliation (General disorders) | 3 | 5
Application site rash (General disorders) | 4 | 3
Application site erythema (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days